CLINICAL TRIAL: NCT04545398
Title: Acute Evidence of Digestive, Metabolic and Nutritional Differences in Beef and Meat- Analogue Meals
Brief Title: Acute Meat and Alternative Intake (PRotEin DIet SatisfacTION Trial 3)
Acronym: PREDITION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Institute for Human Development and Potential (IHDP), Singapore (Other); Massey University (Other); AgResearch (Unknown); The Riddet Institute (Unknown)
Responsible Party: Principal Investigator, Dr Andrea Braakhuis, Principal Investigator, University of Auckland, New Zealand
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 5000927; U1111-1244-9426 (Registry Identifier: Universal Trial Number)
Record Dates: First submitted 2020-05-12; First posted 2020-09-11 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Diet, Healthy; Protein; Disease
Keywords: protein; amino acid; diet; health; meat products; bioavailability
MeSH Terms: conditions — Disease | interventions — Food; Red Meat

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pasture-raised (Experimental): The meal contains grass/pasture fed beef
  Interventions: Other: Food. Beef, Pasture-raised
- Grain-fed (Experimental): The meal contains grain-fed beef
  Interventions: Other: Food. Beef, Grain-fed
- Meat Alternative (Placebo Comparator): The meal contains a meat alternative
  Interventions: Other: Food. Meat alternative
- Lamb (Experimental): The meal contains lamb
  Interventions: Other: Food, Lamb

INTERVENTIONS:
Other: Food. Beef, Pasture-raised — Pasture-raised beef
  Arms: Pasture-raised
Other: Food. Beef, Grain-fed — Grain-fed beef
  Arms: Grain-fed
Other: Food. Meat alternative — Meat alternative
  Arms: Meat Alternative
Other: Food, Lamb — Lamb
  Arms: Lamb

SUMMARY:
Introduction: Protein rich foods that are alternatives to farm-grown meat have received considerable consumer attention. Whilst meat alternatives were once niche food products aimed at vegetarians, they are increasingly marketed to omnivores and "flexitarians", thus contributing to a trend for reductions in red meat intakes [1]. Studies to date have addressed the environmental benefit, plus consumer perceptions and acceptability of meat alternatives [2, 3, 4], yet there is surprisingly a paucity of data compared the nutritional and digestive differences to meat. The aim of this trial is to compare the digestive consequences of pasture-fed and grain-finished, beef versus a plant-based meat analogue blinded meal.

Methods and analyses: Healthy, young (20-34 y) participants will be asked to consume three separate meals in a crossover, blinded investigation followed by five hours of blood testing and questionnaires to assess the digestive consequences of meat and a plant-based meat analogue. The three meals will include either pasture-fed, or grain-finished, or laboratory based protein alternative as a mixed meal, in random order, separated by one week minimum. Plasma samples will be assessed amino acid content, neurotransmitter proteins, chylomicron fatty acid distribution and general health indices.

Ethics and dissemination: The trial has been granted ethical approval by the Ministry of Health, Health and Disability Ethics Committee (Ref: 19/STH/226). All results originating from this study will be submitted for publication in scientific journals and presented at meetings.

DETAILED DESCRIPTION:
Introduction: Red meat consumption contributes important nutrients to the diet, including essential amino acids, long chain and complex lipids, vitamins (including B12) and minerals (including iron and zinc) [5]. While supplying these important nutrients, red meat may contain components which may negate optimal health such as the saturated fat content and nitrates, that are added during processing [5]. The degree to which red meat affects health is likely related to its inherent nutritional profile, the quantity consumed and any processing (e.g. nitrates or cooking techniques). Regardless, the simple notion of a complex whole-food containing single nutrients which are 'good' or 'bad' for health is now considered overly simplistic [6]. For example, to reduce heart disease, nutritional guidelines now suggest an increase in polyunsaturated fats at the expense of saturated fat, rather than a complete reduction of all fats [6].

Alongside the controversy over the health consequences of red meat, recent attention has focused on the possibility of using "plant-based" proteins as an alternative to red meat consumption. The search for meat alternatives has resulted in a sharp increase in the production of novel "plant-based" meat analogues that have been designed to replicate the taste and eating experience of red-meat. To date there are very few studies addressing the nutritional differences between traditional red meat and plant-based meat analogues, and the nutritional differences that arise due to different production systems. Given the nutritional composition of red meat is likely to be influenced by the farming and feeding practices of the animals, production procedures and end-user cooking techniques [7], these differences need to be accounted for in the research design and application.

Aims: To investigate the digestive responses to an acute intake of pasture-fed beef, grain-finished beef, lamb and a plant based meat-analogue consumed as a component of a mixed meal. This study is part of a larger programme to understand the nutritional implications of consuming New Zealand, pasture-fed red meat as part of a balanced diet.

Study Design and Setting: The study is designed as randomised cross-over trial to capture biological difference in postprandial nutrient dynamics. Research subjects will act as their own controls and will consume each meal (pasture raised, grain-fed beef, lamb and a meat alternative meal) on a separate occasion in random order. The study compares exemplars of pasture-fed New Zealand beef, grain-finished New Zealand beef, lamb and a meat analogue. The plant-based meat analogue has been selected on the basis of its macronutrient profile (protein and fat) and appearance in order to that best matches that of meat.

The digestion and metabolism of key nutrients in beef will be measured immediately after the ingestion of a single meal. This experimental setting will also be used to examine some subjective qualities of the meal experience, such as satisfaction score (i.e., liking, satisfaction, enjoyment, satiety, appetite) and gastrointestinal score (i.e., comfort, fullness, bloating, rumbling, flatulence, faecal urgency, diarrhoea).

ELIGIBILITY:
Inclusion Criteria:

* All participants will be required to be omnivores willing to consume both red meat and plant-base alternatives for the purposes of the trial.

Exclusion Criteria:

* Those with chronic health conditions, hyperlipidaemia, obesity (BMI ≥ 30), use of medications (except occasional use of NSAIDs and antihistamines), history of anosmia and ageusia (issues with taste and smell), current dieting or disordered eating pattern and smoking tobacco or recreational drugs will be excluded from participating.
* Participants will be asked to complete an on-line screening which will include the Three-factor Eating Questionnaire-R18 (TFEQ) and a health survey. Participants with a TFEQ score greater than 75% will be excluded from participating on the basis their perception of food is potentially influenced by underlying psychological issues

Ages: 20 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self reported gender is acceptable
Enrollment: 30 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
LCPUFA (18:2 n-6, 18:3 n-3, 20:4 n-6, 20:5 n-3, 22:5 n-3, 22:6 n-3 | Change from baseline to 240-minutes post meal ingestion
  Chylomicron fatty acids, blood test

SECONDARY OUTCOMES:
Fatty acids (14:0, 16:0, 16:1 n-7, 18:0, 18:1 n-9, others) | Change from baseline to 240-minutes post meal ingestion
  Chylomicron fatty acids, blood test
Amino acids/ Neurotransmitters | Change from baseline to 240-minutes post meal ingestion
  blood test
Glucose/ Insulin | Change from baseline to 240-minutes post meal ingestion
  Blood test
Minerals/ Iron | Change from baseline to 240-minutes post meal ingestions
  Blood test
Fullness | Change from baseline to 240-minutes post meal ingestion
  Questionnaire (8 questions), Likert scale, non-directional answers
Digestive Symptoms | Change from baseline to 240-minutes post meal ingestion
  Questionnaire (11 questions), Likert scale, higher score indicative of greater symptoms
Meal Palatability | Difference between intervention meals, 30 minutes post meal
  Questionnaire (5 questions), Likert scale, higher score indicative of greater palatability

CONTACTS AND LOCATIONS:
Overall Officials: Andrea J Braakhuis, PhD, Principal Investigator — The University of Auckland
Locations (1):
- The University of Auckland, Auckland, [other], New Zealand

IPD SHARING:
Plan to Share IPD: Yes
As yet there is no plan but we are open to sharing the data
Supporting Information: Study Protocol, ICF
Time Frame: Pre-recruitment
Access Criteria: The study protocol will be freely available via publication

REFERENCES:
- [Background] 1. Thakur A. Market for Plant-Based Meat Alternatives. Environmental, Health, and Business Opportunities in the New Meat Alternatives Market. IGI Global; 2019: 218-37.
- [Background] Slade P. If you build it, will they eat it? Consumer preferences for plant-based and cultured meat burgers. Appetite. 2018 Jun 1;125:428-437. doi: 10.1016/j.appet.2018.02.030. Epub 2018 Mar 5. PMID 29501683
- [Background] 3. Circus VE, Robison R. Exploring perceptions of sustainable proteins and meat attachment. B Food J. 2019.
- [Background] Keefe LM. #FakeMeat: How big a deal will animal meat analogs ultimately be? Anim Front. 2018 Jul 19;8(3):30-37. doi: 10.1093/af/vfy011. eCollection 2018 Jul. No abstract available. PMID 32002221
- [Background] Ekmekcioglu C, Wallner P, Kundi M, Weisz U, Haas W, Hutter HP. Red meat, diseases, and healthy alternatives: A critical review. Crit Rev Food Sci Nutr. 2018 Jan 22;58(2):247-261. doi: 10.1080/10408398.2016.1158148. Epub 2017 Jun 28. PMID 27128451
- [Background] Forouhi NG, Krauss RM, Taubes G, Willett W. Dietary fat and cardiometabolic health: evidence, controversies, and consensus for guidance. BMJ. 2018 Jun 13;361:k2139. doi: 10.1136/bmj.k2139. PMID 29898882
- [Background] Hicks TM, Knowles SO, Farouk MM. Global Provisioning of Red Meat for Flexitarian Diets. Front Nutr. 2018 Jun 14;5:50. doi: 10.3389/fnut.2018.00050. eCollection 2018. PMID 29963555
- [Derived] Pham T, Morton L, Gillies N, Bermingham E, Knowles S, Cameron-Smith D, Braakhuis AJ. Plasma chylomicron-rich lipidomic and fatty acid profile following a meat or analog meal in healthy males: A randomized controlled trial. Am J Clin Nutr. 2025 Sep;122(3):770-779. doi: 10.1016/j.ajcnut.2025.07.010. Epub 2025 Jul 15. PMID 40675490
- [Derived] Pham T, Knowles S, Bermingham E, Brown J, Hannaford R, Cameron-Smith D, Braakhuis A. Plasma Amino Acid Appearance and Status of Appetite Following a Single Meal of Red Meat or a Plant-Based Meat Analog: A Randomized Crossover Clinical Trial. Curr Dev Nutr. 2022 May 4;6(5):nzac082. doi: 10.1093/cdn/nzac082. eCollection 2022 May. PMID 35669048

DOCUMENTS (2):
  • Study Protocol (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT04545398/Prot_000.pdf
  • Informed Consent Form (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT04545398/ICF_002.pdf